CLINICAL TRIAL: NCT03769519
Title: AdheRence to Inhaled Corticosteroids in Asthma
Acronym: ARICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00100181
Record Dates: First submitted 2018-10-16; First posted 2018-12-07 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Medication Adherence; Asthma
Keywords: health disparities; african american; adult
MeSH Terms: conditions — Medication Adherence; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Group 1) (No Intervention): This group is considered the control group. This group will have scheduled texts and emails for the monthly surveys after the participant completes the baseline questionnaires.
- ARICA Intervention (Group 2) (Experimental): This group is considered the intervention group. Participants in this group will receive weekly texts and emails containing asthma facts and myths. They will also complete monthly surveys and participate in asthma education sessions.
  Interventions: Behavioral: ARICA

INTERVENTIONS:
Behavioral: ARICA — Personalized ARICA (AdheRence to Inhaled Corticosteroids in Asthma) intervention package.
  Arms: ARICA Intervention (Group 2)

SUMMARY:
It is widely recognized that asthma in adult African American patients is a significant health problem, which is partly affected by relatively low inhaled corticosteroid (ICS) adherence rates. The goal of this study is to pilot test an ICS adherence intervention, ARICA, that aims to improve ICS adherence in adult African Americans.

DETAILED DESCRIPTION:
The investigators will evaluate ARICA in Duke primary care clinics to study its feasibility and acceptability using a quasi-experimental pre-post study design. The study will enroll between 32 and 48 adult African Americans with persistent asthma and suboptimal ICS adherence, and their health care providers, to study the use of the intervention and key indicators of the intervention's potential effectiveness.

ELIGIBILITY:
Inclusion Criteria

* At least 18 years of age
* Self-identifying African American
* Self-reported current asthma
* Prescribed an inhaled corticosteroid (alone or combination) for ≥ 1 month
* Presented at a Duke Primary Care clinic visit within the past 3 years or is establishing care at Duke Primary Care
* Follow up Duke Primary Care visit within the next 6 months

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaretta L Riley, MD, Principal Investigator — Duke Un.
Locations (1):
- Duke Un., Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control (Group 1) | ARICA Intervention (Group 2)
Started | 14 | 15
Completed | 14 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Group 1) | ARICA Intervention (Group 2) | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.2) | 47.1 (10.5) | 49.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 14 | 27
  White | 0 | 0 | 0
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
DOSE-Nonadherence (Voils Adherence) [Mean (Standard Deviation); unit: units on a scale] — patients' medication adherence rates based on Voils adherence questionnaire adherence questionnaire. Scored 0-4, higher is more non-adherent
  units on a scale | 1.6 (0.9) | 1.3 (1) | 1.5 (1)
Asthma Control Test [Mean (Standard Deviation); unit: units on a scale] | 14 (5.5) | 16.1 (4) | 15.1 (4.8)
Marks Asthma Related Quality of Life [Mean (Standard Deviation); unit: units on a scale] | 33.2 (17.7) | 23.2 (17.2) | 28 (17.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Experiences With the ARICA Program
Description: Assessment of participants experiences with and perceptions of the ARICA program, as assessed by in-depth semi-structured qualitative interview.
Time Frame: 3 months
Population: Conducted qualitative interview of ARICA Intervention participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Group 1) | ARICA Intervention (Group 2)
Number analyzed (Participants) | 0 | 14
Participants |  | 12

2. Secondary Outcome: Change in Patient Reported Medication Adherence as Measured by the DOSE-Nonadherence (Voils) Questionnaire
Description: patients' medication adherence rates based on Voils adherence questionnaire adherence questionnaire. Difference from baseline to follow up. Scored 0-4, higher is more non-adherent
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control (Group 1) | ARICA Intervention (Group 2)
Number analyzed (Participants) | 14 | 15
score on a scale | 0.685 [-0.0385 to 0.7528] | 0.738 [0.1928 to 1.28]

3. Secondary Outcome: Change in Asthma Control as Measured by the Asthma Control Test
Description: patient reported difference from baseline to follow up. Higher score is better asthma control. Range 5-25.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control (Group 1) | ARICA Intervention (Group 2)
Number analyzed (Participants) | 14 | 14
score on a scale | -2.571 [-5.1902 to 0.0473] | -3.5 [-6.0396 to -0.9604]

4. Secondary Outcome: Change in Asthma-Related Quality of Life as Measured by the Marks Asthma-Related Quality of Life Questionnaire
Description: Patient reported. Difference from baseline to follow up. Range 0-80, higher score means greater impact of asthma on quality of life.
Time Frame: 3 months
Population: Participants who completed the Marks Asthma-Related Quality of Life Questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control (Group 1) | ARICA Intervention (Group 2)
Number analyzed (Participants) | 13 | 13
score on a scale | 5.769 [-1.2527 to 12.7912] | 11.462 [5.5068 to 17.4163]

ADVERSE EVENTS:
Time Frame: Study period, 3 months
Arm/Group | Control (Group 1) | ARICA Intervention (Group 2)
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03769519/Prot_000.pdf